CLINICAL TRIAL: NCT07291414
Title: Patient Engagement in Using the Technology for Self-Tracking Medication Safety Events
Brief Title: A Self-Monitoring Platform for Tracking Medication Safety and Concerns in Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UMCC 2025.050; NCI-2025-08754 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00272763 (Other: University of Michigan); R01HS027846 (AHRQ)
Record Dates: First submitted 2025-12-04; First posted 2025-12-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma; Colorectal Carcinoma; Lung Carcinoma; Malignant Solid Neoplasm; Prostate Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Chromatin Immunoprecipitation Sequencing; Follow-Up Studies; Interviews as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health services research (self-monitoring platform) (Experimental): Patients use the self-monitoring platform to track medication-related safety events and issues at home for 6 months. Patients may receive relevant educational materials and resources via the platform or by email and/or receive follow-up contact from a nurse practitioner as needed over the 6 months. Patients are encouraged to continue using the platform for an additional 6 months after the study period, as desired.
  Interventions: Other: Educational Intervention; Other: Electronic Health Record Review; Procedure: Follow-Up; Other: Internet-Based Intervention; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Receive educational materials and resources
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Electronic Health Record Review — Ancillary studies
Procedure: Follow-Up — Receive follow-up contact
  Other Names: Active Follow-up; Clinical Signs Follow-up; CLSFUP; Follow Up; follow_up; Followed; Followup
Other: Internet-Based Intervention — Use self-monitoring platform
Other: Interview — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the usefulness of a self-monitoring platform for tracking medication safety events and concerns in patients with lung, colorectal, breast, and prostate cancer. Patients receiving oral anticancer agents often encounter challenges in managing complex treatment regimens, potentially life-threatening toxicities, and drug-drug and drug-food interactions at home. To achieve the goal of medication safety, they need to become "vigilant partners" in medication and toxicity self-monitoring, including timely reporting of medication events to clinicians when their care transitions back home. In this study, patients use an online self-monitoring platform to track their experiences or concerns about taking their medications, including their experiences with symptoms. This platform may be a useful way for patients to track problems they have when taking their medications at home and may help them take better care of their health.

ELIGIBILITY:
Inclusion Criteria:

* Participants are adult patients (aged 18 years or older)
* Diagnosed with lung, colorectal, breast, or prostate cancer
* Are currently receiving active cancer treatments
* Are self-managing one or more prescribed cancer medications
* Participants must have access to technology devices (smartphone, tablet, computer) to track their experiences or concerns about medication safety events, or their family members can help them access technology devices to track the events or concerns
* Speaks and reads English or has a support person (family member or friend) who can assist

Exclusion Criteria:

* Can't access technology or do not use technology
* Do not have access to the internet
* Do not speak or read English
* Not permitted to participate by their health care providers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported system usability | Up to 6 months
  Self-reported system usability will be assessed using the 10-item System Usability Scale. Will use descriptive statistics, such as mean and standard deviation for continuous variables, and frequency and percentage for categorical variables.
Perceived usefulness | Up to 6 months
  Qualitative data, including brief interview data will be analyzed and summarized through content analysis.
Ease of use | Up to 6 months
  Qualitative data, including brief interview data will be analyzed and summarized through content analysis.
Attitudes toward use | Up to 6 months
  Qualitative data, including brief interview data will be analyzed and summarized through content analysis.
Intention to use and continuous use of the system over time | Up to 12 months
  Qualitative data, including brief interview data will be analyzed and summarized through content analysis.
Self-reported patient engagement | Up to 6 months
  Self-reported patient engagement will be measured by the 9-item Twente Engagement with Ehealth Technologies Scale (TWEETS), including three dimensions, behavioral engagement, cognitive engagement, and affective engagement. Will use the overall TWEETS score to evaluate patient engagement in this study, rather than analyzing each dimension separately. Will use descriptive statistics, such as mean and standard deviation for continuous variables, and frequency and percentage for categorical variables. Will use repeated measures analysis of variance to assess the changes in mean scores of patient engagement. Univariate associations between baseline personal and clinical factors and patient engagement at each time point will be assessed using correlation analyses (Pearson or Spearman), Chi-square tests, or non-parametric Mann-Whitney U tests, depending on the variable types. Multiple linear regressions will be conducted to assess associations between patient engagement and outcomes.
System usage over time | Up to 12 months
  Will be objectively recorded by the system logs and analyzed using Google Analytics (dashboard only), including parameters like the number of logins, number of tab pages clicked, number of events or concerns self-tracked, and more. Will use descriptive statistics, such as mean and standard deviation for continuous variables, and frequency and percentage for categorical variables.
Patient activation levels | Up to 6 months
  Patient activation levels will be measured by the Short Form of Patient Activation Measure. Will use descriptive statistics, such as mean and standard deviation for continuous variables, and frequency and percentage for categorical variables.
Medication self-management ability | Up to 6 months
  Medication self-management ability will be measured by the Measure of Medication Self-Management. Will use descriptive statistics, such as mean and standard deviation for continuous variables, and frequency and percentage for categorical variables.
Symptom distress | Up to 6 months
  Symptom distress will be measured by the 19-item MD Anderson Symptom Inventory. Will use descriptive statistics, such as mean and standard deviation for continuous variables, and frequency and percentage for categorical variables.
Health related quality of life | Up to 6 months
  Health-related quality of life will be measured by the 27-item Functional Assessment of Cancer Therapy - General. Will use descriptive statistics, such as mean and standard deviation for continuous variables, and frequency and percentage for categorical variables.
Number of emergency room visits | Up to 12 months
  Will be measured by both self-report and chart review. Will use descriptive statistics, such as mean and standard deviation for continuous variables, and frequency and percentage for categorical variables.
Number of hospitalizations | Up to 12 months
  Will be measured by both self-report and chart review. Will use descriptive statistics, such as mean and standard deviation for continuous variables, and frequency and percentage for categorical variables.
User experiences with the system | Up to 6 months
  Participants' user experiences with the system, such as perceived facilitators or barrios to system use, along with their suggestions for system improvement, will be collected through a brief individual interview. Qualitative data, including brief interview data will be analyzed and summarized through content analysis.

SECONDARY OUTCOMES:
Self-tracked, structured medication safety events or concerns | Up to 12 months
  To understand the nature and causes of events and concerns, self-tracked, structured medication safety events or concerns tracking data from the system, such as the number and types of events or concerns self-tracked, will be summarized using descriptive statistics. The free-text tracking data from the system will be analyzed and summarized through content analysis or natural language processing techniques, depending on data volume.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Jiang, Principal Investigator — University of Michigan Rogel Cancer Center; Yang Gong, Principal Investigator — UTHealth Houston McWilliam School of Biomedical Informatics
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No